CLINICAL TRIAL: NCT04674514
Title: Phase Ib / II Open-Label Stduy of APG-2575 Monotherapy or in Combination With Lenalidomide / Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: APG-2575 Monotherapy or in Combination With Lenalidomide/DXMS in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG2575MC101
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Bcl-2 inhibitor; APG-2575
MeSH Terms: conditions — Multiple Myeloma | interventions — Lisaftoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Single agent) (Experimental): Dose escalation APG-2575 at 3 dose levels 3+3 design.
  Interventions: Drug: APG-2575
- Arm B (combo) (Experimental): Dose escalation APG-2575 at 3 dose levels in combination with Rd, 3+3 design.
  Interventions: Drug: APG-2575; Drug: Rd

INTERVENTIONS:
Drug: APG-2575 — APG-2575 orally once daily, every 28 days as a cycle.
Drug: Rd — Lenalidomide administered at a dose of 25 mg orally (PO) on Days 1 through 21 of each 28-day cycle, dexamethasone administered at a dose of 40 mg (or 20 mg for patients>75 years old) on Days 1, 8, 15, and 22 of a repeated 28-day cycle.
  Other Names: Lenalidomide +Dexamethasone
  Arms: Arm B (combo)

SUMMARY:
This is a Phase Ib/II, open-label, multi-center study evaluating the safety, tolerability, efficacy, and PK/ Pharmacodynamics of APG2575 monotherapy or in combination with lenalidomide (R) and dexamethasone (d) in patients with relapsed/refractory (R/R) multiple myeloma (MM). The primary objective is to evaluate the safety and tolerability, identify dose-limiting toxicities (DLT), the maximum tolerated dose (MTD) and the recommended dose (RP2D) of APG-2575 monotherapy or in combination with Rd in Chinese R/R MM patients.

DETAILED DESCRIPTION:
This is a Phase Ib/II, open-label, multi-center study evaluating the safety, tolerability, efficacy, and PK/ Pharmacodynamics of APG2575 monotherapy or in combination with lenalidomide (R) and dexamethasone (d) in patients with relapsed/refractory (R/R) multiple myeloma (MM). The primary objective is to evaluate the safety and tolerability, identify dose-limiting toxicities (DLT), the maximum tolerated dose (MTD) and the recommended dose (RP2D) of APG-2575 monotherapy or in combination with Rd in Chinese R/R MM patients.

This study consists of two arms of APG-2575 single agent (arm A) and APG-2575 in combination with Rd (arm B). All subjects will receive consecutive treatment in 28-day cycles.

All subjects will continue to receive treatment until disease progression, unacceptable toxicities, or other treatment discontinuation criteria fdefined by the protocol. All subjects will complete survival follow up after treatment discontinuation until end of the study, withdrawal of informed consent, loss of follow-up, or death.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age;
2. Life expectancy ≥ 6 months;
3. Eastern Cooperative Oncology Group (ECOG) ≤ 2;
4. Corrected QT interval (QTc) based on Frederica or Bazett formula ≤ ≤450ms (male)，or ≤ 470ms (female);
5. Patients with Relapsed/Refractory MM, previously treated with at least 1 prior line of therapy for MM;
6. Symptomatic MM patients with measurable disease (IMWG 2016);
7. Patients with a history of autologous HSCT must have an adequate bone marrow function and have recovered from any transplant-related toxicity, and meet a minimum of 6 months post-autologous transplant (prior to first dose).
8. Adequate hematologic function without growth factor support
9. Adequate hepatic, renal and coagulation function
10. Male and female subjects of childbearing potential who agree to use highly effective methods of birth control during the period of therapy and for 90 days after the last dose of study drug.
11. Ability to understand and voluntarily sign a written informed consent form before performing any study procedures.
12. Compliance to study procedures.

Exclusion Criteria:

1. monoclonal antibody therapy within 4 weeks prior to first dose; CAR-T therapy within 3 months prior to first dose; or other anti-myeloma therapy within 2 weeks prior to first dose.
2. Only Arm B:intolerance to lenalidomide.
3. Plasma cell leukemia, non-secretory multiple myeloma, Fahrenheit macroglobulinemia, primary amyloidosis, POEMS syndrome.
4. Subjects planning to undergo a stem cell transplant prior to progression of disease on this study, i.e., these subjects should not be enrolled in order to reduce disease burden prior to transplant.
5. Subject has previously received an allogenic stem cell transplant (regardless of timing).
6. Participated in other clinical trial treatments within 14 days before the first dose (calculated from the time of withdrawal from the study treatment).
7. Unable to swallow tablets or malabsorption syndrome, disease significantly affecting gastrointestinal function.
8. Known central nervous system involvement.
9. Failure to have fully recovered (i.e., ≤ Grade 1 toxicity) from the reversible effects of prior treatment.
10. Not recovered from recent surgical procedures based on investigator's discretion. Major surgical procedure within ≤28 days or minor surgical procedure within ≤14 days prior to initiating study treatment, or anticipation of the need for major surgery during the course of the study treatment and 14 days post last treatment, radiotherapy ≤14 days.
11. Unstable angina, myocardial infarction, or coronary revascularization within 180 days prior to the first dose.
12. Active rheumatoid arthritis, active inflammatory bowel disease, or other chronic inflammatory diseases.
13. Active infection need systemic treatment, including HIV antibody positive, HCV Ab or RNA more than ULN, or HBV-DNA more than ULN.
14. Severe uncontrollable medical condition, including, but not limited to, symptomatic congestive heart failure, severe arrhythmias, unstable angina, or a psychiatric disorder that may affect study adherence;
15. Subject has any concurrent or recent malignancy ≤ 5 year prior to registration with the exception of: basal or squamous cell skin cancer and any carcinoma in situ with adequate therapy, or other cancers successfully cured with surgical procedures or drugs ≥ 2 years.
16. Any other condition or circumstance that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.
17. Female patients who are pregnant or breastfeeding.
18. Requires treatment with a strong cytochrome P450 (CYP) 3A4 inhibitor or inducer、strong CYP2C8 inhibitor (except study treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 28 days
  DLT will be defined based on the rate of drug-related grade 3-5 adverse events experienced within the first 28 days of study treatment. These will be assessed via CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Suzhou Yasheng Pharmaceutical Co., Ltd.
Locations (12):
- China (12):
  - Beijing Chao-yang Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Province People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College of Huazhong University of Science ang Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - People's hospital of Jiangsu Province, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affilated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang